CLINICAL TRIAL: NCT00317876
Title: Dose-Finding Study for Cyclophosphamide as Conditioning Regimens for Bone Marrow Transplantation From Related Donors in Patients With Fanconi Anemia
Brief Title: Cyclophosphamide in Treating Patients Who Are Undergoing a Donor Bone Marrow Transplant for Fanconi's Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Hans-Peter Kiem, MD, Fred Hutchinson Cancer Research Center
Masking: None | Purpose: Treatment
Other Study IDs: 1288.00; FHCRC-1288.00; CDR0000481264 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Fanconi Anemia
Keywords: Fanconi anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Cyclophosphamide; Cyclosporine; Methotrexate

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as cyclophosphamide, before a donor bone marrow transplant helps stop the growth of abnormal cells. It also stops the patient's immune system from rejecting the donor's bone marrow. The donated bone marrow stem cells may replace the patient's immune system and help destroy any remaining abnormal cells. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and methotrexate before or after transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of cyclophosphamide in treating patients who are undergoing a donor bone marrow transplant for Fanconi's anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Decrease the conditioning-related toxicity of cyclophosphamide without decreasing the engraftment rate to < 90% in patients undergoing allogeneic bone marrow transplantation for Fanconi's anemia.

OUTLINE: This is a multicenter, dose-finding study of cyclophosphamide.

* Nonmyeloablative conditioning regimen: Patients receive cyclophosphamide IV on days -5 to -2.

Cohorts of 5-10 patients receive decreasing doses of cyclophosphamide until the optimal dose (OD) is determined. The OD is defined as the dose at which ≥ 4 of 5 patients achieve engraftment and < 1 of 10 patients experiences dose-limiting toxicity.

* Allogeneic bone marrow transplantation (BMT): Patients undergo allogeneic BMT on day 0.
* Graft-vs-host-disease (GVHD) prophylaxis: Patients receive cyclosporine orally or IV twice daily beginning on day -1 and continuing until day 49, followed by a taper on days 50-180 in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Fanconi's anemia by chromosome fragility with a diepoxybutane (DEB) or mitomycin C test

  * Hemoglobin ≤ 8.0 g/dL, absolute granulocyte count ≤ 1,000/mm^3, or platelet count ≤ 50,000/mm^3
* No refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, or acute leukemia
* HLA-identical related donor available

PATIENT CHARACTERISTICS:

* Glomerular filtration rate ≥ 30% predicted for age
* No liver disease (e.g., active hepatitis or moderate to severe portal fibrosis/cirrhosis by biopsy)
* No symptomatic cardiac insufficiency or symptomatic arrhythmia
* No other diseases that would severely limit the probability of survival
* No HIV seropositivity
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1998-06; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Conditioning-related toxicity | 100 days post-transplant
Graft rejection | 100 days post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Kiem, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (3):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Universidade Federal do Parana, Curitiba, Paraná, Brazil